CLINICAL TRIAL: NCT03108274
Title: A Three-Part Phase 1 Study to Determine the Potential Drug Interaction Between ACH-0144471 and Midazolam, Fexofenadine and Mycophenolate Mofetil in Healthy Subjects
Brief Title: A Drug Interaction Study Between Danicopan and Midazolam, Fexofenadine, and Mycophenolate Mofetil in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Collaborators: Achillion, a wholly owned subsidiary of Alexion (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: ACH471-010; U1111-1193-2774 (Other: Universal Trial Number (UTN))
Record Dates: First submitted 2017-03-28; First posted 2017-04-11 (Actual); Last update posted 2021-06-24 (Actual); Status verified 2021-06

CONDITIONS: Healthy
Keywords: Danicopan; ALXN2040; ACH-0144471; Midazolam; Fexofenadine; Mycophenolate Mofetil; Drug Interaction; Pharmacokinetics; Factor D Inhibitor; Safety
MeSH Terms: interventions — danicopan; rhoA GTP-Binding Protein; Midazolam; fexofenadine; Mycophenolic Acid

STUDY DESIGN:
Intervention Model Description: Part 1, Part 2, and Part 3 could be conducted concurrently or separately, and the order of the parts could be determined according to the needs of the program.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Part 1: Danicopan and Midazolam (Experimental): Period 1: Participants received a single dose of midazolam.
  Period 2: Participants received multiple doses of danicopan, in addition to coadministration with a single dose of midazolam.
  Scheduled pharmacokinetics (PK) blood samples were collected, with a washout period of at least 3 days between the dose in Period 1 and the first dose in Period 2.
  Interventions: Drug: Danicopan; Drug: Midazolam
- Part 2: Danicopan and Fexofenadine (Experimental): Period 1: Participants received a single dose of fexofenadine.
  Period 2: Participants received multiple doses of danicopan, in addition to coadministration with a single dose of fexofenadine.
  Scheduled PK blood samples were collected, with a washout period of at least 3 days between the dose in Period 1 and the first dose in Period 2.
  Interventions: Drug: Danicopan; Drug: Fexofenadine
- Part 3: Danicopan and MMF (Experimental): Period 1: Participants received a single dose of MMF.
  Period 2: Participants received multiple doses of danicopan, in addition to coadministration with a single dose of MMF.
  Scheduled PK blood samples were collected, with a washout period of at least 3 days between the dose in Period 1 and the first dose in Period 2.
  Interventions: Drug: Danicopan; Drug: Mycophenolate Mofetil

INTERVENTIONS:
Drug: Danicopan — Oral tablet.
  Other Names: ALXN2040; ACH-0144471 (formerly)
Drug: Midazolam — Oral syrup.
  Other Names: Midazolam HCl
  Arms: Part 1: Danicopan and Midazolam
Drug: Fexofenadine — Oral tablet.
  Arms: Part 2: Danicopan and Fexofenadine
Drug: Mycophenolate Mofetil — Oral tablet.
  Arms: Part 3: Danicopan and MMF

SUMMARY:
The purpose of this study was to determine the potential drug interaction between danicopan (ACH-0144471) and midazolam, fexofenadine, and mycophenolate mofetil. This was a 3-part study, with each part being an open-label, fixed-sequence, 2-treatment study in healthy adult participants.

ELIGIBILITY:
Key Inclusion Criteria:

* Healthy was defined as having no clinically relevant abnormalities identified by a detailed medical history, physical examination, blood pressure and heart rate measurements, 12-lead electrocardiogram, and clinical laboratory tests.
* Body mass index of 18.5 to 32 kilograms (kg)/square meter with a minimum body weight of 50 kg.

Key Exclusion Criteria:

* Mentally or legally incapacitated or significant emotional problems.
* Any condition that might interfere with drug absorption.
* History of sensitivity to study medication or other drug allergies.
* Body temperature greater than or equal to 38°Celsius on Day -1 or Day 1 predose; history of febrile illness within 14 days of the first dose.
* Positive urine drug test; current tobacco/nicotine users and smokers; consumption of alcohol within 72 hours of study drug administration.
* Participated in another clinical study within 28 days prior to the first dose.
* Significant laboratory abnormalities.
* Blood donation of more than 500 milliliters within 3 months of the first dose; received a blood transfusion or blood products within 6 months to the first dose.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2017-04-18 (Actual); Primary Completion 2017-06-02 (Actual); Study Completion 2017-06-16 (Actual)

PRIMARY OUTCOMES:
Part 1: Midazolam Area Under The Plasma Concentration-time Curve From Time 0 To The Time Of The Last Observed Non-zero Concentration (AUC0-t) Following Single-dose Midazolam Alone Versus In The Presence of Steady-state Danicopan | Up to 24 hours postdose
Part 1: Midazolam Area Under The Plasma Concentration-time Curve From Time 0 Extrapolated To Infinity (AUC0-inf) Following Single-dose Midazolam Alone Versus In The Presence of Steady-state Danicopan | Up to 24 hours postdose
Part 1: Midazolam Maximum Observed Plasma Concentration (Cmax) Following Single-dose Midazolam Alone Versus In The Presence of Steady-state Danicopan | Up to 24 hours postdose
Part 1: Midazolam Time To Reach Maximum Observed Plasma Concentration (Tmax) Following Single-dose Midazolam Alone Versus In The Presence of Steady-state Danicopan | Up to 24 hours postdose
Part 2: Fexofenadine AUC0-t Following Single-dose Fexofenadine Alone Versus In The Presence of Steady-state Danicopan | Up to 72 hours postdose
Part 2: Fexofenadine AUC0-inf Following Single-dose Fexofenadine Alone Versus In The Presence of Steady-state Danicopan | Up to 72 hours postdose
Part 2: Fexofenadine Cmax Following Single-dose Fexofenadine Alone Versus In The Presence of Steady-state Danicopan | Up to 72 hours postdose
Part 2: Fexofenadine Tmax Following Single-dose Fexofenadine Alone Versus In The Presence of Steady-state Danicopan | Up to 72 hours postdose
Part 3: Mycophenolic Acid (MPA) and Mycophenolic Acid Glucuronide (MPAG) AUC0-t Following Single-dose Mycophenolate Mofetil (MMF) Alone Versus In The Presence of Steady-state Danicopan | Up to 72 hours postdose
Part 3: MPA and MPAG AUC0-inf Following Single-dose MMF Alone Versus In The Presence of Steady-state Danicopan | Up to 72 hours postdose
Part 3: MPA and MPAG Cmax Following Single-dose MMF Alone Versus In The Presence of Steady-state Danicopan | Up to 72 hours postdose
Part 3: MPA and MPAG Tmax Following Single-dose MMF Alone Versus In The Presence of Steady-state Danicopan | Up to 72 hours postdose

SECONDARY OUTCOMES:
Parts 1-3: Participants Experiencing Treatment-emergent Adverse Events | 7 (±1) days following the last dose in Period 2

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Trial Site, Auckland, New Zealand